CLINICAL TRIAL: NCT04158336
Title: A Phase 1 Study of ZN-c3 as a Single Agent in Subjects With Solid Tumors
Brief Title: A Study of ZN-c3 in Participants With Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: K-Group, Beta, Inc., a wholly owned subsidiary of Zentalis Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZN-c3-001
Record Dates: First submitted 2019-11-04; First posted 2019-11-08 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Solid Tumor
Keywords: Uterine Serous Carcinoma; Solid Tumors Harboring Biomarkers Related to DNA Damage Pathways
MeSH Terms: interventions — Drug Evaluation

STUDY DESIGN:
Intervention Model Description: USC Cohort is Parallel Assignment and MOI Cohort is Single Group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Single Agent Dose Escalation (Experimental): Subjects with solid tumors with advanced or metastatic disease who are refractory or ineligible to standard therapy(ies) or for whom no standard therapy is available.
  Interventions: Drug: ZN-c3
- Single Agent Food Effect Cohort (Experimental): Subjects with solid tumors with advanced or metastatic disease who are refractory or ineligible to standard therapy(ies) or for whom no standard therapy is available. This cohort will give subjects the option to continue treatment after PK assessments are completed.
  Interventions: Drug: ZN-c3
- Single Agent Dose Expansion (Experimental): Subjects with histologically confirmed recurrent or persistent USC who have had treatment with at least 1 prior platinum-based chemotherapy regimen for management of advanced or metastatic USC and subjects with locally advanced or metastatic malignancy with one or more relevant biomarkers related to DNA damage pathways.
  Interventions: Drug: ZN-c3

INTERVENTIONS:
Drug: ZN-c3 — ZN-c3 is a study drug
  Other Names: Study Drug

SUMMARY:
This is a Phase 1 open-label, multicenter study of ZN-c3 monotherapy which consists of Dose Escalation, a Food Effect Cohort, and Dose Expansion.

DETAILED DESCRIPTION:
This study will evaluate the safety, tolerability, efficacy, pharmacokinetics (PK) and pharmacodynamics of ZN-c3.

In Dose Escalation, the study will identify the Maximum Tolerated Dose (MTD) of ZN-c3 monotherapy in solid tumors.

The Food Effect cohort sub-study will examine ZN-c3 PK after a single dose and determine the bioavailability of ZN-c3 under fed and fasted conditions.

In Dose Expansion, single agent ZN-c3 will be evaluated at the RP2D in subjects with recurrent or persistent uterine serous carcinoma (USC) or subjects with locally advanced or metastatic solid tumor malignancies harboring biomarkers related to deoxyribonucleic acid (DNA) damage pathways.

ELIGIBILITY:
Major Eligibility Criteria:

1. Age ≥ 18 years or the minimum legal adult age (whichever is greater) at the time of informed consent.
2. Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
3. Adequate hematologic and organ function.
4. Female subjects of childbearing potential and male subjects must agree to use an effective method of contraception and for 6 months and 90 days, respectively, after the last dose of ZN-c3.

Dose Escalation Inclusion Criteria:

1. Subjects must have a solid tumor with advanced or metastatic disease, refractory to standard therapy or for whom no standard therapy is available, or the subject is ineligible for standard therapy(ies).
2. Measurable or evaluable disease per RECIST version 1.1.

Food Effect Cohort Inclusion Criteria:

1. Subjects with solid tumors with advanced or metastatic disease who are refractory or ineligible to standard therapy(ies) or for whom no standard therapy is available.
2. Subjects must have no relevant dietary restrictions, and be willing to consume a high-calorie, high-fat breakfast and other standard meals provided during the study.

Dose Expansion Inclusion Criteria:

1. Measurable disease, defined as at least one lesion that can be accurately measured per RECIST version 1.1 criteria.
2. Recurrent or persistent USC or locally advanced or metastatic malignancy with one or more relevant biomarkers related to deoxyribonucleic acid (DNA) damage pathways.

Major Exclusion Criteria:

1. Prior therapy with ZN-c3 or known hypersensitivity to any drugs similar to ZN-c3 in class or any inactive ingredients present in ZN-c3.
2. Prior therapy with a WEE1 inhibitor.
3. A serious illness or medical condition(s).
4. Unresolved toxicity of Grade >1 attributed to any prior therapies (excluding Grade ≤2 neuropathy, alopecia or skin pigmentation).
5. Pregnant or lactating females (including the cessation of lactation) or females of childbearing potential who have a positive serum pregnancy test within 14 days prior to C1D1.
6. Subjects with active (uncontrolled, metastatic) second malignancies or requiring therapy.
7. 12-lead ECG demonstrating a corrected QT interval using Fridericia's formula (QTcF) of >480 ms, except for subjects with atrioventricular pacemakers or other conditions (e.g., right bundle branch block) that render the QT measurement invalid.
8. History or current evidence of congenital or family history of long QT syndrome or Torsade de Pointes (TdP).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation | Through completion, average of 1 year
  To investigate the safety and tolerability of single agent ZN-c3, including identification of the maximum tolerated dose (MTD)/recommended Phase 2 dose (RP2D), based on the incidence and severity of adverse events (AEs) and dose-limiting toxicities (DLTs) in DLT-evaluable subjects.
Food Effect Cohort | Through completion, approx 6 months
  To characterize and compare the PK (Cmax.) of ZN-c3 following a single dose of ZN-c3 under fed and fasting conditions.
Food Effect Cohort | Through completion, approximately 6 months
  To characterize and compare the PK (Tmax) of ZN-c3 following a single dose of ZN-c3 under fed and fasting conditions.
Food Effect Cohort | Through completion approximately 6 month
  To characterize and compare the PK (AUC0-last,AUC0-∞) of ZN-c3 following a single dose of ZN-c3 under fed and fasting conditions.
Food Effect Cohort | Through completion, approximately 6 mth
  To characterize and compare the PK (T1/2) of ZN-c3 following a single dose of ZN-c3 under fed and fasting conditions.
Dose Expansion | Through completion, approximately 43 month
  To investigate the clinical activity of WEE1 inhibition based on the objective response rate (ORR) as defined by the revised Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

SECONDARY OUTCOMES:
Dose Escalation, Food Effect cohort & Dose Expansion | Through completion
  To obtain preliminary estimates of antitumor efficacy of single agent ZN-c3 based on objective response rate (ORR) as defined by the revised Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Food Effect Cohort | Through completion
  To investigate electrocardiogram intervals (QTc Interval) via Holter monitoring after a single dose of ZN-c3 under fed and fasting conditions.
Dose Escalation, Food Effect cohort and Dose Expansion | Through completion.
  To obtain preliminary estimates of antitumor efficacy of single agent ZN-c3 based on Duration of Response (DOR) as defined by the revised Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Dose Escalation, Food Effect cohort and Dose Expansion | Through completion..
  To obtain preliminary estimates of antitumor efficacy of single agent ZN-c3 based on Progression Free Survival (PFS) as defined by the revised Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Dose Escalation, Food Effect cohort and Dose Expansion | Through completion...
  To obtain preliminary estimates of antitumor efficacy of single agent ZN-c3 based on Clinical Benefit Rate (CBR) defined as complete response, partial response or stable disease according to the revised Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Pultar, MD, Study Director — K-Group Beta, a Zentalis Company
Locations (8):
- United States (8):
  - Site 0102, Tucson, Arizona
  - Site 0167, Newport Beach, California
  - Site 0171, Chicago, Illinois
  - Site 0101, Detroit, Michigan
  - Site 0173, New York, New York
  - Site 0179, Pittsburgh, Pennsylvania
  - Site 0103, Houston, Texas
  - Site 0100, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No